CLINICAL TRIAL: NCT04536571
Title: Vision Stability and Preference for Soft Toric vs. Soft Spherical Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C19-679 (EX-MKTG-115)
Record Dates: First submitted 2020-08-14; First posted 2020-09-02 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Astigmatism; Myopia
MeSH Terms: conditions — Astigmatism; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Contact lens (Experimental): Subjects will be randomized to wear test lenses for 30 minutes, and then cross-over to control lenses.
  Interventions: Device: Test Contact lens; Device: Control Contact lens
- Control Contact lens (Active Comparator): Subjects will be randomized to wear control lenses for 30 minutes, and then cross-over to test lenses.
  Interventions: Device: Test Contact lens; Device: Control Contact lens

INTERVENTIONS:
Device: Test Contact lens — Subjects will be randomized to wear test lenses for 30 minutes, and then cross-over to control lenses.
  Other Names: Soft comfilcon A toric contact lenses
Device: Control Contact lens — Subjects will be randomized to wear control lenses for 30 minutes, and then cross-over to test lenses.
  Other Names: Soft comfilcon A sphere contact lenses

SUMMARY:
The principal hypothesis is to be tested in this work is that vision stability (the primary outcome measure) with a spherical contact lens correction vs. a toric contact lens correction will be the same.

DETAILED DESCRIPTION:
This will be a randomised, subject-masked, crossover, bilateral non-dispensing study, controlled by cross-comparison. Thirty subjects will use each lens type at a single visit in random sequence.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged 18-35 years and have capacity to volunteer.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They are an existing wearer of soft spherical contact lenses in both eyes.
5. They have a spherical component of their spectacle refractive error between

   -0.50DS and -6.50DS in both eyes.
6. They have a cylindrical component of their spectacle refractive error between

   -0.75DC and -1.25DC in both eyes.
7. They can be fitted satisfactorily with both lens types.
8. They own an acceptable pair of spectacles.
9. They agree not to participate in other clinical research for the duration of the study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops (including comfort drops) or ointment on a regular basis.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or breastfeeding.
8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
9. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
10. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD., Principal Investigator — University of Manchester
Locations (1):
- Eurolens Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Contact Lens Then Control Contact Lens: Subjects were randomized to wear test lenses for 30 minutes, and then cross-over to control lenses.
- Control Contact Lens Then Test Lens: Subjects were randomized to wear control lenses for 30 minutes, and then cross-over to test lenses.
Period: First Intervention
Arm/Group | Test Contact Lens Then Control Contact Lens | Control Contact Lens Then Test Lens
Started | 11 | 16
Completed | 11 | 16
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test Contact Lens Then Control Contact Lens | Control Contact Lens Then Test Lens
Started | 11 | 16
Completed | 11 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear either test or control lenses for 30 minutes and then cross-over to the other lens.
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27

OUTCOME MEASURES:

1. Primary Outcome: Vision Stability While Doing Tasks on Mobile Phone
Description: Vision stability was assessed by study subjects while doing tasks on mobile phone using a 0-100 visual analogue scales (0 - Unacceptable. Lens cannot be worn, 100 - Excellent. Unaware of any visual loss)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test Contact Lens: Subjects were randomized to wear test lenses for 30 minutes.
  Test Contact lens: contact lenses.
- Control Contact Lens: Subjects were randomized to wear control lenses for 30 minutes.
  Control Contact lens: contact lenses.
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 27 | 27
units on a scale | 88.37 (10.71) | 85.30 (11.75)

2. Primary Outcome: Vision Stability While Doing Tasks on Desktop
Description: Vision stability was assessed by study subjects while doing tasks on desktop using a 0-100 visual analogue scales (0 - Unacceptable. Lens cannot be worn, 100 - Excellent. Unaware of any visual loss)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 27 | 27
units on a scale | 87.78 (12.04) | 83.41 (15.13)

3. Primary Outcome: Vision Stability While Walking
Description: Vision stability was assessed by study subjects while walking using a 0-100 visual analogue scales (0 - Unacceptable. Lens cannot be worn, 100 - Excellent. Unaware of any visual loss)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test Contact Lens | Control Contact Lens
Number analyzed (Participants) | 27 | 27
units on a scale | 88.15 (14.77) | 82.63 (15.22)

4. Secondary Outcome: Lens Fit for Test Contact Lens
Description: Lens fit was assessed for lens rotation after 10 minutes for toric fit. Lens mislocation from optimal position was measured in 0°, 1-5°, 6-10°, 11-15°, 16-20°, More than 20°.
Time Frame: 10 minutes
Measure: Number; unit: Number of Lenses
Groups:
- Test Contact Lens - Right Eye; Test Contact Lens - Left Eye: Subjects were randomized to wear test lenses - Toric Lens rotation was recorded at 10 minutes after dispense.
Arm/Group | Test Contact Lens - Right Eye | Test Contact Lens - Left Eye
Number analyzed (Participants) | 27 | 27
Number of Lenses
  0° | 8 | 9
  1-5° | 16 | 17
  6-10° | 2 | 0
  11-15° | 1 | 1
  16-20° | 0 | 0
  More than 20° | 0 | 0

5. Secondary Outcome: Lens Fit
Description: Lens fit was assessed as either 'acceptable' or 'not acceptable' for standard fit by study investigator.
Time Frame: 30 minutes
Measure: Number; unit: participants
Groups:
- Test Contact Lens: Subjects were randomized to wear test contact lenses for 30 minutes.
  Test Contact lens
- Control Contact Lenses: Subjects were randomized to wear control lenses for 30 minutes.
Arm/Group | Test Contact Lens | Control Contact Lenses
Number analyzed (Participants) | 27 | 27
participants
  Acceptable | 27 | 27
  Not Acceptable | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline till 30 minutes on each study lenses, a total of 1 hour.
Groups:
- Test Contact Lens: Subjects were randomized to wear test lenses for 30 minutes, and then cross-over to control lenses.
  Test Contact lens: contact lenses.
- Control Contact Lens: Subjects were randomized to wear control lenses for 30 minutes, and then cross-over to test lenses.
  Control Contact lens: contact lenses.
Arm/Group | Test Contact Lens | Control Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT04536571/Prot_SAP_000.pdf